CLINICAL TRIAL: NCT01425346
Title: Freedom Meditech ClearPath DS-120 Clinical Study Protocol FM2-002-CTP
Brief Title: ClearPath DS-120 Clinical Study Protocol
Status: Completed | Type: Observational
Sponsor: Freedom Meditech (Industry)
Responsible Party: Sponsor
Other Study IDs: FM2-002-CTP
Record Dates: First submitted 2011-08-24; First posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Ophthalmic, Healthy Eyes
Keywords: Ophthalmic, healthy eye, fluorescence, lens

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Healthy: Normal, healthy males and females between the ages of 21 and 70 with healthy eyes as determined by a standard ophthalmic examination.

SUMMARY:
The goal of this study is to measure lens fluorescence in normal subjects at various chronological ages that could serves as a guide to clinicians in determining changes in eye health. A measure of lens fluorescence can be used by clinicians as an indication of degenerative changes occurring in the lens of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Persons between the ages of twenty-one (21) and seventy (70). Best efforts shall be made to include as many patients as possible between the ages of thirty-five (35) and sixty (60).
* Subject must be able to read or understand and give informed consent.
* Pass the medical health history and comprehensive ophthalmic examination (which is determined by the investigator if the test subject has a normal ophthalmic examination and is in overall good health). Ophthalmic examination includes a clinical evaluation of the subject's eyes and a complete manifest refraction producing a best aided visual acuity of <20/40.

Exclusion Criteria:

* Subject has had the crystalline lens removed from the study eye or has had the crystalline lens removed and replaced with an intraocular lens (IOL) implant in the left eye.
* Subject has been clinically diagnosed with cataracts in the study eye.
* Subject has had a fluorescence angiogram within the last six months.
* Subject has undergone a treatment using photodynamic drugs within the last year.
* Subject has Type I or II diabetes or is not deemed healthy from Demographic and Health Questionnaire or the comprehensive eye exam.
* Subject was fit with contact lens within the last 30 days.
* Subject has ocular surface (dry eye) disease.
* Subject is unable to cooperate with or understand clinical instructions.
* Subject is unable to complete test sequence

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, normal subject population with healthy eyes as determined by standard comprehensive ophthalmic examination.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Lens fluorescence | Day 1
  evaluate the ability of the ClearPath DS-120 instrument to measure the fluorescence and scattering responses of the human crystalline lens in a normal subject population with healthy eyes (as determined by standard comprehensive ophthalmic examination).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen W. Lum, O.D., Principal Investigator — San Diego Optometry Practice
Locations (1):
- San Diego Optometry Practice, San Diego, California, United States